CLINICAL TRIAL: NCT05408949
Title: Effectiveness of Single Exercise Into Pain Program Versus Shoulder Symptom Modification Procedure With Early Tendon Loading, Heavy Slow Resistance Exercise in Patients With Rotator Cuff-related Shoulder Pain: a Randomised Controlled Trial
Brief Title: Comparison of SEP Exercises Versus SSMP With Tendon Loading & Resistance Exercise in Shoulder Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB/COHS/STD/06/Jan-2022; IRB/COHS/STD/06/Jan-2022 (Other: Gulf Medical University)
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Subacromial Pain Syndrome
Keywords: Subacromial pain syndrome, Rotator cuff tendinopathy

STUDY DESIGN:
Intervention Model Description: Randomized control trial 13-weeks parallel non-inferiority study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double (participant, investigators) blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEP+FR (Experimental): - Single exercises program (SEP) is considered to be harmless, valid and has a valuable prescription as initial rehabilitation program. studies showed an immediate analgesic relief and increase in muscle strength after preforming single heavy-load isometric training program
  Interventions: Behavioral: Single exercise into pain (SEP) program; Behavioral: Functional Rehabilitation Program
- SSMP+ETL+HSR+FR Group (Active Comparator): * The Shoulder Symptom Modification Procedure (SSMP) consists of applying several mechanical techniques and applied when the patient moves or performs a specific activity. This procedure is designed to address the symptoms and improve range of motion by identifying mechanical changes.
  * Heavy slow resistance (HSR) training is an alternative from traditional exercise physiotherapy, by emphasizing on heavy weights and slow repetition. HSR training includes repetitive gradual and slow contraction of the muscle during concentric, isometric and eccentric phases against a heavy weight
  * Early controlled and progressive tendon loading (EPTL) in rehabilitation practice is suggested to show a high and definite impact on healing and recovery of the tendon
  Interventions: Behavioral: Shoulder Symptom Modification Procedure (SSMP); Behavioral: Functional Rehabilitation Program; Behavioral: EPTL; Behavioral: HSR

INTERVENTIONS:
Behavioral: Single exercise into pain (SEP) program — * Baseline assessment & commencement of treatment: Resisted isometric shoulder abduction into pain (or lateral rotation or flexion into pain) against a wall, or Resisted shoulder abduction from 0 to 30° using moderate resistance from Theraband ( Prescribed High intensity loading to the tendon (85-90% iMVC) applied in 5 repetitions with a 45 secoud hold (3 times per week)).
  * Initial follow-up & progression: Resisted shoulder abduction into pain from 80 to 120° using light weight (Prescribed High intensity loading to the tendon (85-90% iMVC) applied in 5 repetitions with a 45 secoud hold (3 times per week)).
  * Second follow-up & progression: eccentric shoulder abduction into pain from 80 to 120° with progressively increasing repetition and weight, e.g. heavy Theraband or dumbbell.
  * Final assessment to identify any non-resolved functional limitations and progress eccentric exercises into pain as required
  * Functional rehabilitation program
  Arms: SEP+FR
Behavioral: Shoulder Symptom Modification Procedure (SSMP) — [1] Finger on the sternum,[2A] Scapula modification [3] 'Humeral head' modification [4] Isometric (most painful movement) Heavy slow resistance (HSR): start from the mid-range and pain-free
  Arms: SSMP+ETL+HSR+FR Group
Behavioral: Functional Rehabilitation Program — Mostly targetted into exercise such as multi-stage pushing, pulling, lifting and carrying, throwing, kinetic chain exercises and aerobics. FR involved (i). Weight-shifting activities to enhance dynamic joint stability[18] .(ii). Proprioceptive neuromuscular facilitation exercises to stimulating stretch receptors located on the muscle or tendon units [18]. Using resistive tubing exercises in a functional position using PNF patterns; diagonal pattern 1: flexion, abduction, external rotation (10-15 repetition 2-3 sets). (iii) Plyometric exercise: (A) throwing motions; (B) push-up (10-15 repetition 2-3 sets) . (iv). Table slide (10-15 repetition 2-3 sets).
Behavioral: EPTL — In EPTL it involves eccentric training in Full range (with dumbbells 15-10 RM) of Internal and external rotation at scapular plane elevation (0-45) degree and Flexion, Abduction, in full range (5 repetitions with a 45 second hold at slow speed) to target the series elastic component of the muscle .
  Arms: SSMP+ETL+HSR+FR Group
Behavioral: HSR — In HSR it involves eccentric training in mid-range of motion (with dumbbells 15-10 RM) targeting the contractile component of the muscles and improving mechanical strength. Additionally, when there is 90% pain reduction on NPRS functional rehabilitation program start and they follow the same program as Group A.
  Arms: SSMP+ETL+HSR+FR Group

SUMMARY:
Shoulder pain is one of the most prevalent and disabling musculoskeletal condition. A new diagnostic terminology used to describe shoulder pain is rotator cuff-related shoulder pain (RCRSP), as histological findings were similar in many of shoulder condition such as; subacromial impingement syndrome, subacromial pain syndrome and rotator cuff tendinopathy The objectives was to find the effectiveness of single exercise into pain program versus Shoulder Symptom Modification Procedure (SSMP) with early tendon loading, Heavy Slow Resistance exercise in patients with rotator cuff-related shoulder pain.

The investigators will conducted a randomized clinical trail in out patient physiotherapy department at Thumbay hospitals Ajman, in patients with rotator cuff-related shoulder pain . After meeting the inclusion criteria, participants were randomized into Single exercises into pain program (SEP) (intervention group) or Shoulder Symptom Modification Procedure (SSMP) with early tendon loading, Heavy Slow Resistance exercise program (control group).

A 13 weeks of outpatient musculoskeletal rehabilitation sessions consisting of 3 sessions per week will provided to both the groups. Intervention group will receive single exercises into pain by preforming resisted isometric shoulder abduction with TheraBand and progressed to functional rehabilitation, whereas control group will receive a combination of shoulder symptom modification to control the pain, early tendon loading to target the series elastic component of the muscle and heavy slow resistance program to target contractile component of the muscles and improve mechanical strength followed by functional rehabilitation.

The investigators will measured Shoulder Pain and Disability Index (SPADI), Numerical Pain Rating Scales (NPRS), and Digital Wall (D-WALL) H-Sport Quality Of Life at the baseline assessment, 6th weeks and 13th weeks

DETAILED DESCRIPTION:
The Shoulder Symptom Modification Procedure (SSMP) is a series of mechanical techniques that are applied while the patient performs the activity or movement, with the aim of identifying a mechanical change that will alleviate and treat the symptoms and improve range of motion. This process involves identifying the movement, posture, or activity that reduces the patient's symptoms. SSMP is designed to identify a positive effect on symptoms by providing changes in position of the glenohumeral or scapulothoracic joints or thoracic spine. Besides, SSMP perhaps impact the symptoms related with RCRSP by altering rotator cuff muscle-tendon tension, changing the anatomical structure, and releasing the neuromodulation. Using Shoulder Symptom Modification Procedure (SSMP) can inspect the effect of thoracic spine posture, scapula posture in three different anatomical planes, and position of humeral head on shoulder joint symptoms. Moreover, it provides immediate direction for selecting one or more methods among the four mechanical techniques for treating RCRSP. The main goal of SSMP to treat, decrease symptoms and/or improving function and movement.

Heavy slow resistance (HSR) training program includes repetitive gradual and slow contraction of the muscle during concentric, isometric and eccentric phases against a heavy weight, i.e., 1RM. In previous studies it was proven that the HSR training program used for a plantar fasciopathy was found to have superior results than stretching. Demonstrating Heavy Slow Resistance in eccentric form will target the contractile component of the muscles and improve mechanical strength. Besides HSR training is an alternative from traditional exercise physiotherapy, by emphasizing on heavy weights and slow reptation. Without sufficient power the muscle and tendons will have poor strength and endurance. A suggestion of static, sustain load with 5 reptation and 45 second hold, repeated 2-3 times per week will provide a beneficial outcome. Only one recent study showed a 15% increase in abduction due to adding heavy load eccentric training for individuals with unilateral subacromial impingement.

Administration of early controlled and progressive tendon loading (EPTL) in rehabilitation practice is suggested to show a high and definite impact on healing and recovery of the tendon. In addition, there are various benefits related to EPTL, new evidence showed it help accelerates healing, alleviate joint restriction, and reduce the risk of re-tearing. Moreover, it has been stated that load exercises for mid-tendon or at the insertion sites of the Achilles tendon provide a better clinical outcome in any parts of the tendon. Besides, preforming isometrics in mid-range can reduce the pain in tendinopathy rehab progression.

Furthermore, single exercises into pain (SEP) program is considered to be harmless, valid and has a valuable prescription as initial rehabilitation program. A recent study discussed the tendinopathy in lower limbs showed an immediate analgesic relief and increase in muscle strength after preforming single heavy-load isometric training program. Pain can be better used for navigate the symptom management to foster recovery. A "Traffic Light Pain Control graph" where a score of 3 out of 10 pain level is a good area to practice the exercise. In addition, a score of 4 out of 10 isn't harmful or can cause any damage. Although pain level should be tolerable and isn't increasing the next day. Additionally in Reactive tendinopathy/early tendon disrepair level, the load management helps the matrix of the tendon to resume a more normal structure. However, the clinical effectiveness of SEP on shoulder conditions is still sparce.

Daily functional rehabilitation (FR) is needed for the individual with RCRSP to provide self-independence after the initial phases of physiotherapy. In the functional activity, daily living or sporting activities of the individuals are incorporated in an exercise form to train and facilitate pain free and efficient daily movement contingencies. a daily functional rehabilitation is needed to avoid any future harm, along with restoring the individuals to their best physical fitness statues. Core stabilization, postural alignment kinetic chain, scapular position, range of motion, pain and cardiovascular training are the main stay of current functional rehabilitation regimes. However little or no research studying the efficacy of functional training programs on the improvement of clinical outcomes of RCRSP. The fundamental reason for this research is that rotator cuff-related shoulder pain can cause a major complication with substantial implication on well-being. A study needed to be conducted to fuel the necessary advances in a newly approaches discovered recently to address and evaluate the clinical effectiveness of above approaches.

Comparing these interventions may provide vital clues for shoulder rehabilitation in the management of RCRSP

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 to 60 years old
2. Rotator Cuff tendinitis, tendinopathy and impingement syndrome
3. Acute and chronic conditions
4. Self-reported pain or symptoms localized around the shoulder, and not referred below the elbow
5. Willing and able to participate, provide consent process

Exclusion Criteria:

1. Inability to communicate or provide informed consent.
2. History of unstable fracture/dislocation in upper extremities with shoulder instabilities
3. Referred pain to shoulder from other area
4. Adhesive capsulitis
5. Any surgical history on shoulder and neck

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | Day 1 of enrollment session and end day of 6th week, change in SPADI scores are assessed
  SPADI is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. The change in SPADI scores are assessed.
  Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.
Numerical Pain Rating Scales (NPRS) | Day 1 of enrollment session and end day of 6th week, change in NPRS scores are assessed
  NPRS will be used to identify the intensity of the participants pain at the baseline, 6th week, and 13th week at rest, activity, night, maximum and the results will be reported. In NPRS, the participants are asked to draw a circle on the number between zero to ten. Zero will represent "no pain at all", ten will represents "'the worst pain ever possible. The change is pain scores are assessed
The Shoulder Pain and Disability Index (SPADI) | End of 6th week and end of 13th week, change in SPADI scores are assessed
  SPADI is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. The change in SPADI scores are assessed.
  Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.
Numerical Pain Rating Scales (NPRS) | End of 6th week and end of 13th week, change in NPRS scores are assessed
  NPRS will be used to identify the intensity of the participants pain at the baseline, 6th week, and 13th week at rest, activity, night, maximum and the results will be reported. In NPRS, the participants are asked to draw a circle on the number between zero to ten. Zero will represent "no pain at all", ten will represents "'the worst pain ever possible. The change is pain scores are assessed.

SECONDARY OUTCOMES:
Digital Wall (D-WALL) H-Sport | Time Frame: From the start of treatment i.e., Day 1, Base line assessment, 6th week and 13th week of therapy session
  A 3D camera which will provide an immediate biofeedback degrees measurement
Patient Global Impression of Change (PGIC) | Time Frame: From the start of treatment i.e., Day 1 and 13th week of therapy session
  Patient Global Impression of Change (PGIC) used and provided a score to help for a better understanding of the patient's progress and overall changes in their symptoms to the healthcare provider. PGIC provides a patient's evaluation of overall improvement on a 7-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ramprasad Muthukrishnan, Ph.D, Principal Investigator — College of Health Sciences, Department of Physiotherapy
Locations (2):
- United Arab Emirates (2):
  - Gulf Medical University, Thumbay Physical Therapy and Rehabiliation Hospital, Thumbay University Hospital, Ajman
  - Gulf Medical University, Ajman

IPD SHARING:
Plan to Share IPD: No
Data will be stored for an year after dissemination of results